CLINICAL TRIAL: NCT06560047
Title: Danish Evaluation of Early Catheter Ablation for Atrial Fibrillation in Patients With Heart Failure - The DanAblate-HF Trial
Brief Title: Danish Evaluation of Early Catheter Ablation for Atrial Fibrillation in Patients With Heart Failure
Acronym: DanAblate-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Zealand University Hospital (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Sam Riahi, Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20240001; F2024-063 (Other: Region NordJylland)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Heart failure; Atrial fibrillation; Catheter ablation; Treatment; Outcome
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: The DanAblate-HF trial is a pragmatic, investigator-initiated, prospective, multicenter, open-labeled, randomized, controlled trial. Patients will be randomized 1:1 to either early catheter ablation or standard treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter Ablation (Other): Patients randomized to the intervention will undergo early catheter ablation with pulmonary vein isolation as treatment for AF. Catheter ablation should be conducted within 6 weeks of randomization.
  Interventions: Procedure: Catheter ablation
- Standard treatment (No Intervention): Patients randomized to standard treatment will receive standard guideline directed treatment for AF and HF. Treatment will be initiated at the baseline visit and further clinical follow-up will be conducted at the patients local hospital. Patient will be treated with either rhythm (excluding catheter ablation) or rate control. The choice of treatment strategy will be at the discretion of the treating physician according to current guideline recommendations. If rate control is chosen, patients should have a resting heart rate < 110 beats per minutes. Rate control can be obtained by medical treatment with digoxin, beta-blockers and if needed amiodarone, in combination or as single treatment. Rhythm control will be conducted through cardioversion and/or medical treatment with amiodarone. Catheter ablation will not be part of the treatment choices in the standard treatment arm.

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation with pulmonary vein isolation will be the study intervention. Patients randomized to the intervention arm will undergo catheter ablation within six weeks of randomization. In the waiting-time for ablation, patients will receive standard treatment for AF and HF, as per current guideline recommendations. Catheter ablation will be performed at one of six high-volume ablation centers in Denmark. Mode of catheter ablation will be at the discretion of the operator. Radiofrequency ablation, cryo-balloon ablation and pulsed-field ablation will be utilized. The treating physician should ensure successful pulmonary vein isolation after ablation with either post-procedural mapping or pacing, as per current standards. Only pulmonary vein isolation will be performed during the ablation procedure.
  Arms: Catheter Ablation

SUMMARY:
The DanAblate-HF trial will investigate whether early catheter ablation treatment for atrial fibrillation in patients with heart failure is superior to standard treatment.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia in patients with heart failure (HF), with rates ranging between 20-65%, depending on age, severity of HF, subtypes of HF and duration of HF. The two conditions have an intricate and often overlapping pathophysiology, with each condition leading to development of the other, as well as progression of disease. Studies have shown that the presence of AF in HF patients is associated with increased morbidity and mortality, deterioration in HF, exacerbated HF symptoms, and reduced quality of life. The optimal treatment of AF in the presence of HF remains unknown. Currently, there is a pull towards catheter ablation as first-line therapy for AF in HF patients. However, there is no solid scientific evidence to support this approach. Furthermore, it is unknown whether early rhythm control by catheter ablation in HF patients is beneficial.

The investigators aim to conduct a pragmatic, randomized clinical trial designed to evaluate the efficacy and safety of early catheter ablation for AF in patients with HF compared with standard treatment.

Eligible patients with HF and AF will be prospectively screened from all Danish hospitals and randomized 1:1 to early catheter ablation with pulmonary vein isolation (within 6 weeks) or standard guideline directed treatment for AF. Patients with reversible causes for AF, conditions that preclude the use of catheter ablation or previous catheter ablation for AF will be excluded from the study. Randomization and follow-up will be conducted at six specialized sites in Denmark. There will be one scheduled on-site 12-months follow-up visit after randomization. All clinical follow-up will be conducted at the patient's local hospital, according to standard practice and out of trial setting. Information regarding hospital visits/admissions, events, adverse events, changes in medication, cross-over, heart rhythm and rate, and results of relevant blood-work will be ascertained through systematic patient chart-review at pre-specified time-points. The results from this trial will mold future treatment of AF in HF patients. The investigators hypothesize that early catheter ablation reduces the risk of HF hospitalizations and mortality when compared with standard treatment, thereby significantly improving the clinical prognosis for patients with HF and AF.

ELIGIBILITY:
Inclusion Criteria:

1. HF patients with AF within the past 12 months

   HF is defined as all of the below (all must apply)
   * Clinically assessed Heart Failure with Reduced Ejection Fraction (HFrEF)
   * An indication for initiation or ongoing guideline directed medical therapy for HFrEF, according to current Heart Failure guidelines
   * LVEF < 50% at any point during the past 12 months

   AF is defined as one or more of the following:

   A. Symptomatic AF, documented by ECG, Holter of CIED

   B. Asymptomatic AF with one or more of the following:
   * Clinical indication for rhythm or rate control (documented by ECG, telemetry, Holter, CIED)
   * ≥2 ECG detected AF episodes within 3 months (on separate dates)
   * Holter detected AF with a continuous duration of more than 6 hours
   * CIED detected AF with continuous duration >24 hours
2. 18 years ≤ Age <80 years
3. Optimal medical therapy for HFrEF or planned/current uptitration in guideline directed medical therapy for HFrEF
4. Treatment with anticoagulation for stroke prevention, initiated according to guidelines for treatment of AF

Exclusion Criteria:

1. Life-expectancy < 1 year
2. BMI > 40
3. Contraindications or unacceptable side effects to rate limiting drugs AND amiodarone
4. LA size (indexed for BSA) > 60 ml/m2 (volume) on echo within the last year
5. Documented persistent/permanent AF > 1 year
6. Previous AF ablation/surgery
7. Reversible causes of AF (including, but not limited to, infection within 14 days, untreated thyroid disease, surgery)
8. Severe valvular disease
9. Acute myocardial infarction, cardiothoracic surgery or stroke within the past 3 months
10. Planned cardiothoracic surgery
11. Listed for heart transplant
12. Contraindications for anticoagulation therapy or catheter ablation
13. Severe kidney disease (CKD≥5)
14. Pregnancy
15. Patient unwilling to try medical therapy for AF
16. Patient unwilling/unable to give informed consent for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1616 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2039-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to hospitalization for worsening HF or cardiovascular death | From baseline to study completion, with a minimum of 1 year
  The primary outcome of the trial is defined as the time from randomization to the composite of one the following, whichever comes first
  * Hospitalization for worsening HF
  * Cardiovascular (CV) mortality
  Hospitalization for worsening HF will be defined as hospital admission primarily for HF (as deemed so by the event adjudication committee) with a duration of at least 24 hours and requiring intensification of diuretic treatment.
  CV mortality will be defined as all deaths resulting from one or more of the following: HF, stroke, acute myocardial infarction, CV procedural deaths, CV hemorrhage, arrythmia, sudden cardiac death, death due to other CV causes and death of undetermined cause.

SECONDARY OUTCOMES:
Time to cardiovascular death | From baseline to study completion, with a minimum of 1 year
  Time from randomization to cardiovascular death. Cardiovascular death will be defined as in the primary endpoint.
Time to all-cause mortality | From baseline to study completion, with a minimum of 1 year
  Time from randomization to all-cause mortality
Time to first heart failure hospitalization | From baseline to study completion, with a minimum of 1 year
  Time from randomization to first hospitalization for heart failure, as defined in the primary endpoint
Time to first-time AF hospitalization | From baseline to study completion, with a minimum of 1 year
  Time from randomization to first hospitalization for AF
Time to primary outcome stratified by age | From baseline to study completion, with a minimum of 1 year
  Time from randomization to trial primary outcome stratified by median age at baseline
Time to primary outcome stratified by sex | From baseline to study completion, with a minimum of 1 year
  Time from randomization to trial primary outcome stratified by sex
Time to primary outcome stratified by symptomatic and asymptomatic AF | From baseline to study completion, with a minimum of 1 year
  Time from randomization to trial primary outcome stratified by whether patients have symptomatic or asymptomatic AF at baseline
Time to primary outcome stratified by paroxysmal or persistent AF | From baseline to study completion, with a minimum of 1 year
  Time from randomization to trial primary outcome stratified by paroxysmal or persistent AF at baseline
Time to primary outcome stratified by left ventricular ejection fraction (LVEF) | From baseline to study completion, with a minimum of 1 year
  Time from randomization to trial primary outcome stratified by LVEF <=40% and LVEF>40% at baseline
Change in Quality of Life | From baseline to 12 months
  Change in Quality of Life will be assessed through Kansas City Cardiomyopathy Questionnaire (KCCQ-23) at baseline and 12 months.
  The KCCQ-23 quantifies physical function/limitations, symptoms, quality of life, social function/limitations and self-efficacy. Scores are generated for each domain and scaled from 0 to 100, with higher scores reflecting better health outcome.
Change in self-assessed health | From baseline to 12 months
  Change in self-assessed health will be assessed through short form-36 (SF-36) questionnaire at baseline and 12 months.
  The SF-36 questionnaire consists of 8 domains: Physical functioning, limitions due to physical health, limitations due to emotional problems, fatigue, emotional well-being, social functioning, general bodily pain and general health. Each domain is scored from 0 to 100, with higher scores reflecting better self-assessed health.
Change in New York Heart Association (NYHA) class | From baseline to 12 months
  Change in NYHA class assessed at baseline and 12 months visit
Change in European Heart Rhythm Association score of atrial fibrillation (EHRA class) | From baseline to 12 months
  Change in EHRA class assessed at baseline and 12 months visit

OTHER OUTCOMES:
Change in LVEF | From baseline to 12 months
  Change in LVEF assessed at baseline echocardiography and 12 months echocardiography
Change in left ventricular (LV) volume | From baseline to 12 months
  Change in LV volume assessed at baseline echocardiography and 12 months echocardiography
Change in left atrial (LA) volume | From baseline to 12 months
  Change in LA volume assessed at baseline echocardiography and 12 months echocardiography
Change in NT-pro-BNP | From baseline to 12 months
  Change in NT-pro-BNP assessed at baseline and 12 month
Time to hospitalization or death due to stroke | From baseline to study completion, with a minimum of 1 year
  Time from randomization to hospitalization or death due to stroke
Cumulative heart failure hospitalization | From baseline to study completion, with a minimum of 1 year
  Total cumulative number (first and recurrent) of hospitalization for heart failure from randomization to study completion.
Cumulative hospitalizations for AF | From baseline to study completion, with a minimum of 1 year
  Total cumulative number (first and recurrent) of hospitalization for AF from randomization to study completion.
Time to first-time all-cause hospitalization | From baseline to study completion, with a minimum of 1 year
  Time from randomization to first all-cause hospitalization
Cumulative all-cause hospitalizations | From baseline to study completion, with a minimum of 1 year
  Total cumulative number (first and recurrent) of all-cause hospitalization from randomization to study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Riahi, MD, PhD, Principal Investigator — Department of Cardiology, Aalborg Univeristy Hospital
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Department of Cardiology, Aalborg
  - Aarhus University Hospital, Aarhus
  - Department of Cardiology, Rigshospitalet, Copenhagen
  - Department of Cardiology, Herlev-Gentofte University Hospital, Hellerup
  - Department of Cardiology, Odense University Hospital, Odense
  - Department of Cardiology, Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No